CLINICAL TRIAL: NCT01216696
Title: Phase II Trial of Ipilimumab in Patients With Advanced Melanoma and Spontaneous Preexisting Immune Response to NY-ESO-1
Brief Title: Ipilimumab in Patients With Advanced Melanoma and Spontaneous Preexisting Immune Response to NY-ESO-1
Acronym: CTLA4 NY-ESO-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2009-11-02-53
Record Dates: First submitted 2010-09-27; First posted 2010-10-07 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Melanoma
Keywords: ipilimumab; melanoma; NY-ESO-1
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Intervention Details:
  Drug: ipilimumab
  Eligible patients will receive 10 mg/kg ipilimumab every 3 weeks during a 10-week induction period, followed by a radiological assessment in week 12. Patients with clinical benefit will continue with an ipilimumab administration every 3 months starting at week 24 up to week 48 until the end of the study or until disease progression, toxicities requiring discontinuation , withdrawal of consent,pregnancy, death or lost to follow up whichever occurs first.
  Interventions: Drug: ipilimumab

INTERVENTIONS:
Drug: ipilimumab — Eligible patients will receive 10 mg/kg ipilimumab every 3 weeks during a 10-week induction period, followed by a radiological assessment in week 12. Patients with clinical benefit will continue with an ipilimumab administration every 3 months starting at week 24 up to week 48 until the end of the study or until disease progression, toxicities requiring discontinuation , withdrawal of consent,pregnancy, death or lost to follow up whichever occurs first.

SUMMARY:
This is an Open-label, single-arm, phase II study of ipilimumab in patients with spontaneous preexisting immune response to NY-ESO-1.

Preclinical data suggest, that CTLA-4 blockade enhances polyfunctional T cell responses in patients with melanoma. Thus patients with immunological response to NY-ESO-1 might benefit from an anti CTLA-4 treatment.

Eligible patients will receive 10 mg/kg ipilimumab every 3 weeks during a 10-week induction period, followed by a radiological assessment in week 12. Patients with clinical benefit (partial response, complete response or stable disease according to the immune-related response criteria) will continue with an ipilimumab administration every 3 months starting at week 24 up to week 48 until the end of the study or until disease progression,toxicities requiring discontinuation

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of malignant melanoma; unresectable Stage III melanoma or Stage IV melanoma; Measurable/evaluable disease (as per mWHO criteria), within 28 days before first dose of study drug;
* Preexisting spontaneous immune response to NY-ESO-1, defined by positive results in ELISA above a prespecified cut-off value.
* Previously treated or untreated metastatic melanoma. The previous treatment must have been finished at least 28 days before the first ipilimumab administration. Patients must have recovered from any acute toxicity associated with prior therapy
* Life expectancy of ≥ 16 weeks;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Men and women, ages 18 and above.
* Ability of subject to understand character and individual consequences of the clinical trial
* Required values for initial laboratory tests:

  * WBC ≥ 2000/μL
  * ANC ≥ 1000/μL
  * Platelets ≥ 100 x 103/μL
  * Hemoglobin ≥ 9 g/dL (may be transfused)
  * Creatinine ≤ 2 x ULN
  * AST/ALT ≤ 2.5 x ULN for subjects without liver metastasis≤ 5 x ULN for subjects with liver metastasis
  * Bilirubin ≤ 2.0 x ULN
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study

Exclusion Criteria:

* Brain Metastasis, unless previously treated, off steroids for at least 4 weeks and considered to be stable (eg, no progression of the treated lesion);
* Primary ocular or mucosal melanoma
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been adequately treated, such as basal or squamous cell skin cancer.
* Autoimmune disease: subjects with a documented history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease are excluded from this study as are subjects with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]). Subjects with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome) are excluded from this study
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Previous participation with a NY-ESO 1 derived vaccination study.
* Inadequate hematologic function defined by an absolute neutrophil count (ANC) < 1,000/mm3, a platelet count < 100,000/mm3, or a hemoglobin level < 9 g/dL;
* Inadequate hepatic function defined by a total bilirubin level > 2.0 x ULN except subjects with Gilbert's Syndrome, who must have a total bilirubin < 3.0 ULN. AST and ALT levels ≥ 2.5 times the ULN, or ≥ 5 times the ULN if liver metastases are present;
* Inadequate renal function defined by a serum creatinine level ≥ 2.0 times the ULN, or inadequate creatinine clearance defined as less than 50 mL/min;
* Positive tests for HIV, Hepatitis B, and Hepatitis C. If positive results are not indicative of true active or chronic infection, the patient can enter the study after discussion and agreement with the investigator and the Medical Monitor.
* Chronic use of immunosuppressants and/or systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses).
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 4 weeks prior to or after any dose of ipilimumab);
* Prior treatment with a CD137 agonist, ipilimumab or other CTLA-4 inhibitor.
* Prisoners or subjects who are involuntarily incarcerated
* Participation in other clinical trials or observation period of competing trials, respectively during the last 30 days before the first application of the investigational agent .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate according to immune-related response criteria | 1 year
  To determine the efficacy of ipilimumab in patients with stage III and stage IV malignant melanoma and spontaneous preexisting immune response to NY-ESO-1.

SECONDARY OUTCOMES:
Progression-free survival according to the immune-related response criteria | 1 year
  To document progression-free survival (PFS) in patients with evaluable or measurable disease after receiving ipilimumab according to the immune-related response criteria (irRC),
Overall Survival at 12 months | 1 year
  To document overall-survival (OS) rate at 12 months after the first study treatment in patients receiving ipilimumab.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year
  To assess the safety profile of ipilimumab in patients with malignant melanoma stage III and IV and spontaneous preexisting immune response to NY-ESO-1.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Jäger, MD, Principal Investigator — NCT Heidelberg, Dep. of Medical Oncology
Locations (1):
- NCT, Dep. of Medical Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Haag GM, Zoernig I, Hassel JC, Halama N, Dick J, Lang N, Podola L, Funk J, Ziegelmeier C, Juenger S, Bucur M, Umansky L, Falk CS, Freitag A, Karapanagiotou-Schenkel I, Beckhove P, Enk A, Jaeger D. Phase II trial of ipilimumab in melanoma patients with preexisting humoural immune response to NY-ESO-1. Eur J Cancer. 2018 Feb;90:122-129. doi: 10.1016/j.ejca.2017.12.001. Epub 2018 Jan 5. PMID 29306769